CLINICAL TRIAL: NCT00348127
Title: A Singapore Pilot Study To Evaluate The Efficacy Of A Computerized System For The Vision Improvement Of People With Low Myopia
Brief Title: A Singapore Pilot Study to Assess Neurovision in Treatment of Low Myopia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Singapore National Eye Centre (Other Government)
Collaborators: Singapore Eye Research Institute (Other); NeuroVision (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R313/06/2003
Record Dates: First submitted 2006-07-03; First posted 2006-07-04 (Estimated); Last update posted 2010-06-24 (Estimated); Status verified 2010-01

CONDITIONS: Myopia
Keywords: Neurovision; Myopia Therapy
MeSH Terms: conditions — Myopia

INTERVENTIONS:
Device: Neurovision

SUMMARY:
To assess how well and safe is Neurovision technology in improving the vision of people with low myopia in Singapore

DETAILED DESCRIPTION:
The eye care industry has focused a majority of its resources on solving problems associated with the ocular or "front end" of the visual system. These investments have led to exciting technology advances, such as intraocular lenses (IOLs) and Laser Vision Correction (LVC) as well as in the development of contact lenses and improved eyewear.

NeuroVision's innovative Neural Vision Correction (NVC) technology has been developed through research focused solely on optimizing performance of the neural or "back end" of the visual system. NeuroVision's technology is distinguished from other products in this space by the Company's expert understanding of how the brain processes vision, its reliance on scientific and clinical research

It is the result of two decades of research by Dr. Uri Polat, founder, who has dedicated 20 years of scientific and clinical research to understanding how the brain processes visual information, how neural activity is related to visual perception, and how visual processing interacts with other neural systems. His work has been published in leading scientific journals and is widely cited by the scientific community.

NeuroVision's NVC vision correction technology is a non-invasive, patient-specific treatment based on visual stimulation and facilitation of neural connections responsible for vision.

The technology has been clinically proven in the treatment of adult amblyopia ("lazy eye"), which until now has been considered untreatable. The Company has received FDA 510(k) marketing clearance indicating NVC for the treatment of adult amblyopia in patients 9 years or older in the US. The Company also received Medical CE-Mark to market its Amblyopia and Low-Myopia products in the EU. Company products are also approved for use in Israel by the Israeli Ministry of Health - Device License Authority.

This study was a prospective non-controlled preliminary clinical study as a prelude to a randomized clinical trial, evaluating the efficacy and safety of NeuroVision NVC correction technology in improving visual acuity and contrast sensitivity function.

ELIGIBILITY:
Inclusion Criteria:

1. The subject's cycloplegic spherical equivalence in the worst eye does not exceed -1.5 DS and the astigmatism does not exceed 0.50 DC.
2. The subject's refractive status is stable, with no increase beyond 0.5D in sphere or cylinder over the last six months.
3. The subject's age is between 17-55 years.
4. The subject's uncorrected visual acuity 0.7 LogMar
5. The subject's best corrected visual acuity 0.05 LogMar
6. The subject is cognitively intact and is able to follow multiple step instructions.
7. The subject is able and willing to attend all study sessions and visits at the required frequency:

   1. The total number of treatments is individual, approximately 30.
   2. The required pace for the treatment sessions is at least 3 sessions per week.
   3. No foreseen interruptions longer than 2 weeks during the treatment course.
8. Subject (or subject's parent/legal guardian if subject is less than 21 years of age at study entry) agrees to sign the Informed Consent Form (See Appendix D)

Exclusion Criteria:

1. The subject suffers from any other eye disease(s) or other causes for the reduced visual acuity, aside from myopia and/or astigmatism.
2. The subject suffers from myopia-related visual complications resulting in visual loss, including myopic macular degeneration, myopic cataract and previous or pre-existing myopic retinal detachment.
3. The subject is suffering from Diabetes Mellitus.
4. The subject has previously undergone a refractive surgery procedure in either eye.
5. The subject is or may be pregnant.
6. The subject has an activity limitation due to medical disorders (including migraines, seizure disorders, etc.), medications, or emotional status that might potentially impair the subject's ability to perform the treatment.

Ages: 15 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 2003-03; Primary Completion 2004-10 (Actual); Study Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
Manifest Subjective and Objective refraction
Cycloplegic Objective refraction
Accommodation amplitude
Distance visual acuity (Uncorrected Visual Acuity - UCVA, and BCVA)
Near visual acuity
Contrast sensitivity (corrected and uncorrected)
Visual Evoked Potential (VEP) and Multifocal VEP

CONTACTS AND LOCATIONS:
Overall Officials: Donald Tan, FRCS, Principal Investigator — Singapore Eye Research Institute
Locations (1):
- Singapore Eye Research Institute, Singapore, Singapore

REFERENCES:
- [Background] Polat U, Ma-Naim T, Belkin M, Sagi D. Improving vision in adult amblyopia by perceptual learning. Proc Natl Acad Sci U S A. 2004 Apr 27;101(17):6692-7. doi: 10.1073/pnas.0401200101. Epub 2004 Apr 19. PMID 15096608
- [Background] Polat U, Mizobe K, Pettet MW, Kasamatsu T, Norcia AM. Collinear stimuli regulate visual responses depending on cell's contrast threshold. Nature. 1998 Feb 5;391(6667):580-4. doi: 10.1038/35372. PMID 9468134
- [Background] Levi DM, Polat U, Hu YS. Improvement in Vernier acuity in adults with amblyopia. Practice makes better. Invest Ophthalmol Vis Sci. 1997 Jul;38(8):1493-510. PMID 9224277
- [Background] Polat U, Norcia AM. Neurophysiological evidence for contrast dependent long-range facilitation and suppression in the human visual cortex. Vision Res. 1996 Jul;36(14):2099-109. doi: 10.1016/0042-6989(95)00281-2. PMID 8776476
- [Background] Sagi D, Tanne D. Perceptual learning: learning to see. Curr Opin Neurobiol. 1994 Apr;4(2):195-9. doi: 10.1016/0959-4388(94)90072-8. PMID 8038576
- [Background] Polat U, Sagi D. Spatial interactions in human vision: from near to far via experience-dependent cascades of connections. Proc Natl Acad Sci U S A. 1994 Feb 15;91(4):1206-9. doi: 10.1073/pnas.91.4.1206. PMID 8108388
- [Background] Polat U, Sagi D. Lateral interactions between spatial channels: suppression and facilitation revealed by lateral masking experiments. Vision Res. 1993 May;33(7):993-9. doi: 10.1016/0042-6989(93)90081-7. PMID 8506641
- [Background] Levi DM, Polat U. Neural plasticity in adults with amblyopia. Proc Natl Acad Sci U S A. 1996 Jun 25;93(13):6830-4. doi: 10.1073/pnas.93.13.6830. PMID 8692904
- See also: Singapore Eye Research Institute — http://www.seri.com.sg/
- See also: Singapore National Eye Centre Website — http://www.snec.com.sg/Pages/home.aspx